CLINICAL TRIAL: NCT06576778
Title: The Impact of Provisionalization Using Fiber-Reinforced Composite on the Quality of Life and Bone Height Changes in Maxillary Implant Supported Arches Restored by Final PEKKTON Frameworks: A Randomized Controlled Trial
Brief Title: The Effect of Fiber-Reinforced Composites on Quality of Life and Bone Height in Maxillary Implant Arches
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Haydi Hesham Mohamed Issa, principle investigator ( assistant lecturer of prosthodontics), Cairo University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 3 1 24
Record Dates: First submitted 2024-08-19; First posted 2024-08-29 (Actual); Last update posted 2024-08-29 (Actual); Status verified 2024-08

CONDITIONS: Edentulous Alveolar Ridge

STUDY DESIGN:
Intervention Model Description: Group I, (control): patients obtained an Implant-supported, full arch maxillary definitive prosthesis utilizing 6 implants, for constructing PEKKTON framework without provisionalization.
  Group II, (intervention): Patients obtained an Implant-supported full arch maxillary provisional prosthesis protocol utilizing 6 implants for constructing a resin glass fiber composite framework followed by a definitive PEKKTON framework.
Who Masked: Outcomes Assessor
Masking Description: The study is based on different technical procedures of framework fabrication. Since these differences are visible, the operator and the patients involved in the study cannot be blinded. But the outcome assessor and the statistician will be blinded.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- No Provisional Prosthesis (PEKKTON as Definitive Framework) (Active Comparator): Implant-supported full arch maxillary prosthesis utilising 6 implants, for constructing PEKKTON framework without provisionalization.
  Interventions: Procedure: PROVSIONALIZATION
- Glass Fiber Reinforced Composite Framework for Provisionalization Then PEKKTON Framework (Experimental): Implant-supported full arch maxillary prosthesis utilising 6 implants, then Glass fiber composite as a temporary framework followed by PEKKTON definitive framework.
  Interventions: Procedure: PROVSIONALIZATION

INTERVENTIONS:
Procedure: PROVSIONALIZATION — glass fiber composite as a temporary framework followed by PEKKTON definitive framework.

SUMMARY:
The aim of this study is assessing the effect of provisionalization with a glass fiber composite framework on patients' quality of life and bone height changes before the insertion of a definitive PEKKTON framework of screw-retained maxillary implant-supported prosthesis at a one-year follow-up period.

DETAILED DESCRIPTION:
1. Patient grouping:

   Group I, (control): patients obtained an Implant-supported, full arch maxillary definitive prosthesis utilizing 6 implants, for constructing PEKKTON framework without provisionalization.

   Group II, (intervention): Patients obtained an Implant-supported full arch maxillary provisional prosthesis protocol utilizing 6 implants for constructing a resin glass fiber composite framework followed by a definitive PEKKTON framework.
2. Preparation of a scan appliance:

   * The patient's denture will be used as a scan appliance by the addition of radiopaque material to act as radiopaque markers over the polished surfaces of the prosthesis in a staggered pattern at different levels to the occlusal plane on the buccal, labial, and palatal flanges of the denture.
   * Double scan protocol will be used in our study in which a cone beam conventional tomography (CBCT) images will be produced for each case. The first scan will be taken for the maxilla while the patient is wearing the maxillary denture with the radiopaque markers and biting over cotton rolls, the other scan is for the modified maxillary denture.
   * Computer software (BlueSky Bio) was used to overlap the two scans on each other where the final file contained reformatted images in 3D bone model, and 3D radiographic modified denture guide model to construct the surgical guide.
3. Virtual planning, surgical guide fabrication, and Implant placement

   * The implant planning will be done using the BlueSky Bio software. The scan of the maxillary denture will be superimposed over that of the maxillary arch scan, using points over the radiopaque marker as alignment points, for proper orientation of the scan appliance.
   * 6 Implant planning ( 3.7x12 for anterior segment and 4x10 for the posterior segment) will be placed in areas with high bone quality and quantity of bone and will be distributed according to AP spread.
   * A surgical guide will be planned and then the 3D virtual guide will be exported as STL file to the 3D printing machine. The surgical guide will be fixed in place using three fixation screws; with an adequate distance from the planned implant drilling sites, two screws placed in the buccal shelf area on both sides and one screw in the midline to achieve a tripoding position.
   * The 3D surgical guide will be provided with metal sleeves corresponding to the virtually planned drilling sites with the precise depth, angulation, mesiodistal and buccolingual positioning of each implant as planned during the computer simulation for accurate placement of the implants' osteotomies. The osteotomies will be drilled, and implants will be inserted.
   * The Multi-unit abutments will be placed over the dental implants, the denture will be relieved and picked up with soft liner.
   * All patients will be instructed about oral hygiene measures, a soft diet for 4 weeks after surgery, and antimicrobial prophylaxes (amoxicillin 500mg twice daily for 5 days starting 1 hour before surgery). Postsurgical analgesic treatment will be performed with ibuprofen 600mg twice daily.
4. Prosthetic procedures:

After 1 Month:

Group I (control gp): patients obtained an Implant-supported, full arch maxillary prosthesis utilizing 6 implants, for constructing PEKKTON framework without provisionalization.

A. Digital impressions Scan bodies will be tightened onto the multi-unit abutments and an intraoral digital impression will be made using an IOS system after one month of implant insertion.

B. Verification jigs fabrication (digitally) The milled PMMA jig will be constructed and checked for passive seating on implants by verifying proper contact at the PMMA jig interface and the multi-unit abutments.

C. Framework fabrication:

* The (PEKKTON) frameworks and teeth will be digitally designed according to implant location, crown height space, occlusion, and opposing dentition with the help of scan appliance wax up.
* The frameworks will be milled with the final material (PEKKTON) and teeth will be printed with temporary material (PMMA).
* First, the passive fit will be checked between frameworks and multi-unit abutments, and the occlusion of printed teeth by PMMA will be checked and tried intra-orally.

Accordingly, if the try-in is accepted, the assigned material (PMMA) will be milled and assembled to the framework.

Group two (intervention gp): will be rehabilitated by using a glass fiber composite as a temporary framework followed by PEKKTON definitive framework.

Framework fabrication:

* The glass fiber composite framework and PMMA teeth will be digitally designed according to implant location, crown height space, occlusion, and opposing complete denture with the help of scan appliance wax up.
* The framework will be placed over the multi-unit abutments intraorally, picked up on cylinder. The occlusion of printed teeth by PMMA will be checked and then cemented with the framework. Then the whole assembly will be removed from patient mouth.
* After one month, the printed composite framework with the printed PMMA teeth will be screwed intraorally.
* After four months of temporization, the definitive PEKKTON will be re-milled from the same scan and delivered to the patients with the milled teeth.
* These frameworks will be milled, the passive fit will be checked between frameworks and multi-unit abutments, and the occlusion of printed teeth by PMMA will be checked and tried intra-orally. If the try-in is accepted, the assigned material (PMMA) will be milled and assembled to the framework.

ELIGIBILITY:
Inclusion Criteria:

* • Completely edentulous patients with Angle's Class I maxillomandibular relationship

  * Age ranges from 40 to 65 years old.
  * Adequate zone of keratinized attached mucosa (≥ 8mm) over the maxillary crest.
  * Absence of any medical disorder that could complicate the surgical phase or affect osseointegration.
  * The patient must have enough bone height for implants, a minimum length of bone
  * 12 mm, and a minimum diameter of bone 6 mm.
  * Patients with good oral hygiene.
  * Adequate inter arch space for screw-retained prosthesis.
  * Absence of any intra-oral pathological condition.

Exclusion Criteria:

* • Patients with recent extraction (less than three months).

  * Patients with an inflamed ridge or candida infection
  * Patients with the flabby ridge.
  * Para functional habits.
  * Cancer patients receiving chemotherapy and/or radiotherapy.
  * Patients with uncontrolled diabetes, assessed by measuring glycosylated hemoglobin (HbA1c ≥ 7)
  * Potentially uncooperative patients who are not willing to go through the proposed interventions.
  * Moderate-to-heavy daily smokers (more than ten per day)

Ages: 40 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 8 (Estimated)
Dates: Start 2024-09 (Estimated); Primary Completion 2025-09 (Estimated); Study Completion 2025-11 (Estimated)

PRIMARY OUTCOMES:
Oral health related to quality of life | 1 year
  A translated form from a validated questionnaire will be used to address the Egyptian population; all patients have to answer the same questionnaire. Each answer will be given a score from 0 to 4 where the lesser the score the better the quality of life, data will be collected, and privacy will be ensured.

SECONDARY OUTCOMES:
Bone height changes assessments | 1 year
  Digital periapical radiographs (Digora System) at the time of implant loading, three months, six-months, one year post-operatively will be done utilizing periapical radiographs following the standardized long cone paralleling technique and evaluated. For further standardization, the same x-ray machine will be used at 8 milliamperes and 70 kilovolts for 0.6 seconds with a focal film distance of 35 cm.
  Marginal bone height changes around the implants will be evaluated using the measurement software system supplied with the Digora radiographs system.

CONTACTS AND LOCATIONS:
Overall Officials: Haydi Issa, PhD, Principal Investigator — faculty of dentistry, Cairo University, Egypt

IPD SHARING:
Plan to Share IPD: No